CLINICAL TRIAL: NCT00352248
Title: Randomized Controlled Trial of Acupuncture Versus Sham Acupuncture in Autistic Spectrum Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9608944339555027
Record Dates: First submitted 2006-07-13; First posted 2006-07-14 (Estimated); Last update posted 2006-07-14 (Estimated); Status verified 1999-07

CONDITIONS: Autistic Disorder; Autism
Keywords: Alternative Medicine (AM); Traditional Chinese Medicine; Tongue Acupuncture; Autistic Spectrum Disorder; Autism; Children
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

INTERVENTIONS:
Procedure: Tongue Acupuncture (Procedure)

SUMMARY:
We aim to study the efficacy of Acupuncture versus sham acupuncture in children with ASD.

DETAILED DESCRIPTION:
In Traditional Chinese Medicine (TCM) philosophy, the approach to Autistic Spectrum Disorder (ASD) is a holistic one. The objective is to study the efficacy of a short intensive course of Acupuncture versus sham acupuncture in improving the overall functional status of children with autism. A single-blind randomized control trial was conducted in 50 children. These children were randomly assigned to Treatment group with Tongue Acupuncture (40 sessions over 8 weeks) or Control group (Sham Tongue Acupuncture to non-acupoints in the tongue).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with diagnosis of autism made according to the criteria of the 4th edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) and Autism Diagnostic Interview-Revised and with a score for Childhood Autism Rating Scale (CARS) greater than 30.

Exclusion Criteria:

* Children with associated neurological disorders and epilepsy.

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50

PRIMARY OUTCOMES:
Griffiths Mental Developmental Scale (GMDS) was conducted before (at Week 0) and after (at Week 9) acupuncture.
Ritvo-Freeman Real Life Scale (RFRLS) was conducted before (at Week 0) and after (at Week 9) acupuncture.
Reynell Language Developmental Scale (RLDS) was conducted before (at Week 0) and after (at Week 9) acupuncture.
Symbolic Play Test (SPT) was conducted before (at Week 0) and after (at Week 9) acupuncture.
Functional Independence Measure for children (WeeFIM) was conducted before (at Week 0) and after (at Week 9) acupuncture.

CONTACTS AND LOCATIONS:
Overall Officials: Wong Virginia, Principal Investigator — The University of Hong Kong
Locations (1):
- Duchess of Kent of Children Hospital, Hong Kong, Hong Kong